CLINICAL TRIAL: NCT06285214
Title: Multicenter, Randomized, Double-blind Placebo-controlled, Crossover Study to Investigate Effects of V117957 in Female Subjects With Interstitial Cystitis/Bladder Pain Syndrome
Brief Title: Study of V117957 in Interstitial Cystitis/Bladder Pain Syndrome
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Imbrium Therapeutics (Industry)
Collaborators: Purdue Pharma LP (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: OAG1050
Record Dates: First submitted 2024-02-22; First posted 2024-02-29 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2025-02

CONDITIONS: Interstitial Cystitis/Bladder Pain Syndrome
MeSH Terms: conditions — Cystitis, Interstitial

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- V117957 (Experimental)
  Interventions: Drug: V117957
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: V117957 — V117957 1 mg - 1 tablet taken orally at bedtime.
  Arms: V117957
Drug: Placebo — Placebo to match V117957 tablets - 1 tablet taken orally at bedtime.
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability and efficacy of V117957 in subjects with interstitial cystitis/bladder pain syndrome, compared to placebo.

ELIGIBILITY:
Key Inclusion Criteria include:

1. Female, age ≥18 years and capable of voiding independently. Able to comply with acceptable methods of contraception.
2. Diagnosis of IC/BPS or meets criteria for IC/BPS as defined by the American Urology Association as "an unpleasant sensation (pain, pressure, discomfort) perceived to be related to the urinary bladder, associated with lower urinary tract symptoms for more than six weeks duration, in the absence of infection or other identifiable causes".
3. Subject has Bladder Pain/Interstitial Cystitis Symptom Scale (BPIC-SS) total score of ≥19 and worst bladder pain/discomfort sub-score of ≥4 to ≤9.
4. Has undergone evaluation to rule out other conditions that cause bladder pain/discomfort. Any microscopic or gross hematuria that has not been evaluated in the past 12 months will require appropriate clinical evaluation to determine study eligibility.

Key Exclusion Criteria include:

1. Pelvic floor tenderness in the absence of bladder tenderness on physical examination by primary investigator.
2. Urinary tract infection (UTI) within the past 30 days, or history of recurrent UTI.
3. Hematuria determined to be associated with bladder malignancy or other significant pathology.
4. Had surgical procedure at any time that affected bladder function.
5. Received intravesical therapy or had bladder hydrodistension, fulguration, botulinum toxin, or triamcinolone bladder injection, percutaneous nerve stimulation. A subject receiving such treatment(s) prior to screening is eligible if in the opinion of the investigator the procedure/ treatment resulted in no notable or enduring effect and subject continues to exhibit stable symptomology.
6. Has current or history of clinically significant kidney disease or abnormal kidney function, or nephrolithiasis.

Other protocol-specific inclusion and exclusion criteria may apply.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2022-05-26 (Actual); Primary Completion 2025-01-28 (Actual); Study Completion 2025-01-28 (Actual)

PRIMARY OUTCOMES:
Change from baseline for bladder pain/discomfort scores over last 12 hours (morning and evening). | Baseline, Weeks 2, 4, 6, 8, and 9
  Each evening and morning the subject will respond to the question "Please indicate the worst bladder pain/discomfort you have had overnight/over the day" using an 11-point NRS that ranges from 0= "no bladder pain/discomfort" to 10= "as bad as you can imagine bladder pain/discomfort."

SECONDARY OUTCOMES:
Change from baseline in mean number of micturitions per 12 hours (morning and evening) | Baseline, Weeks 2, 4, 6, 8, and 9
Change from baseline in Patient Perception of Intensity of Urgency Scale (PPIUS) | Baseline, Weeks 2, 4, 6, 8, and 9
  The PPIUS is a 5-point scale designed for measurement of both urinary urgency and urge incontinence. Subjects are asked to indicate their micturition episode type (urinated= passed urine in the toilet, incontinence= involuntary release of urine) and then rate the episode urgency on a 5-point scale (0= no urgency, 1= mild urgency, 2= moderate urgency, 3= severe urgency, 4= urge incontinence).
Change from baseline in Bladder Pain / Interstitial Cystitis Symptom Score (BPIC-SS) | Baseline, Weeks 2, 4, 6, 8, and 9
  The BPIC-SS contains 8 questions concerning bladder pain over the previous 7 days. Questions 1-5 assess how often subject urinated because of pain, needed to urinate just after a previous urination, urinated to avoid pain, had pressure in their bladder, and had pain in their bladder, are rated on a 5-point scale from 1= "never" to 5= "always." Question 6 and 7 assess how bothered the subject was by frequent urination during daytime and during the night, rated on a 5-point scale from 1= "not at all" to 5= "a great deal." Question 8 assesses subject's worst bladder pain in past 7 days, rated on an 11-point NRS with range 0= "no bladder pain" to 10= "worst possible bladder pain." The BPIC-SS total score is the sum of the individual question scores and range from 0 to 38 with higher scores indicating a worse situation; a score of ≥19 may represent moderate/severe disease activity.
Change from baseline in O'Leary-Sant Interstitial Cystitis Symptom Index (ICSI) | Baseline, Weeks 2, 4, 6, 8, and 9
  The ICSI contains 4 questions that measure urgency and frequency of urination, nighttime urination, and pain or burning. Each question is rated using a 6- or 5-point scale. Total scores range from 0 to 21.
Change from baseline in O'Leary-Sant Interstitial Cystitis Problem Index (ICPI) | Baseline, Weeks 2, 4, 6, 8, and 9
  The ICPI contains 4 questions that assesses and how much of a problem the symptoms cause for the subject. Each question is rated using a 5-point scale. Total scores range from 0 to 16.
Change from baseline in Subject Global Response Assessment (SGRA) | Baseline, Weeks 2, 4, 6, 8, and 9
  The SGRA is a self-rated balanced measure of subject's clinical condition relative to baseline. There is 1 question: "Compared to your last visit, how would you rate your overall overactive bladder symptoms now?" A 7-point rating scale is used: 1= "markedly worse", 2= "moderately worse", 3= "slightly worse", 4= "no change", 5= "slightly improved", 6= "moderately improved" or 7= "markedly improved".
Change from baseline in Symptom Impact Sleep Questionnaire (SISQ) | Baseline, Weeks 2, 4, 6, 8, and 9
  The SISQ contains 2 questions that assess the quality of sleep and the impact of the subject's symptoms of IC/BPS on sleep and is to be completed each morning.

CONTACTS AND LOCATIONS:
Locations (24):
- United States (24):
  - Urology Centers of Alabama, PC, Homewood, Alabama
  - Urological Associates of Southern Arizona, Tucson, Arizona
  - Applied Research Center of Arkansas, Little Rock, Arkansas
  - Investigational Site, Escondido, California
  - Urology Group of Southern California, Los Angeles, California
  - Hope Clinical Research, LLC, Los Angeles, California
  - Tri Valley Urology Medical Group, Murrieta, California
  - Accel Research Sites, DeLand, Florida
  - Accel Research Site - Neurostudies, Decatur, Georgia
  - Providea Health Partners LLC, Evergreen Park, Illinois
  - Otrimed Clinical Research, Edgewood, Kentucky
  - Southern Clinical Research Associates, Metairie, Louisiana
  - Ochsner Louisiana State University Health Shreveport - Regional University, Shreveport, Louisiana
  - Chesapeake Urology Research Associates, Owings Mills, Maryland
  - Boston Clinical Trials, Boston, Massachusetts
  - Bay State Clinical Trials, Inc., Watertown, Massachusetts
  - Revive Research Institute, Inc, Dearborn Heights, Michigan
  - CentraCare - Urology Clinic, Sartell, Minnesota
  - Adult & Pediatric Urology P.C., Omaha, Nebraska
  - AccuMed Research Associates, Garden City, New York
  - Manhattan Medical Research Practice, New York, New York
  - Unified Women's Clinical Research-Lyndhurst Clinical Research, Winston-Salem, North Carolina
  - MetroHealth System, Cleveland, Ohio
  - MidLantic Urology, Bala-Cynwyd, Pennsylvania

IPD SHARING:
Plan to Share IPD: No